CLINICAL TRIAL: NCT00824629
Title: Direct Transfer vs Previous Cervical Canalization Transfer ("Afterloading"): Randomized Clinical Trial.
Brief Title: Embryo Transfer: Direct Versus Afterloading Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Buenaventura Coroleu, Departamento de Obstetricia, Ginecologia y Reproducción
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEX001
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2009-08

CONDITIONS: Infertility
Keywords: Embryo transfer; IVF; Ultrasound embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Afterloading embryo transfer procedure
  Interventions: Procedure: Afterloading embryo transfer procedure
- 2 (Active Comparator): Direct embryo transfer procedure
  Interventions: Procedure: Direct embryo transfer procedure

INTERVENTIONS:
Procedure: Afterloading embryo transfer procedure — Afterloading embryo transfer procedure
  Arms: 1
Procedure: Direct embryo transfer procedure — Direct embryo transfer procedure
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate two types of embryo transfer procedure.

The investigators will compare direct embryo transfer against afterloading embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Patients in IVF/CICSI program
* Transfer day:2 or 3 after ovum pick-up

Exclusion Criteria:

* None

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 8 weeks after embryo transfer

SECONDARY OUTCOMES:
Difficulty of embryo transfer | During embryo transfer procedure
Duration of embryo transfer | During embryo transfer procedure

CONTACTS AND LOCATIONS:
Overall Officials: Buenaventura Coroleu, PhD., MD., Study Director — Departamento de Obstetricia, Ginecologia y Reproduccion , Institut Universitari Dexeus
Locations (1):
- Departamento de Obstetricia Ginecologia y Reproducción. Institut Universitari Dexeus, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Coroleu B, Carreras O, Veiga A, Martell A, Martinez F, Belil I, Hereter L, Barri PN. Embryo transfer under ultrasound guidance improves pregnancy rates after in-vitro fertilization. Hum Reprod. 2000 Mar;15(3):616-20. doi: 10.1093/humrep/15.3.616. PMID 10686207
- [Background] Coroleu B, Barri PN, Carreras O, Martinez F, Parriego M, Hereter L, Parera N, Veiga A, Balasch J. The influence of the depth of embryo replacement into the uterine cavity on implantation rates after IVF: a controlled, ultrasound-guided study. Hum Reprod. 2002 Feb;17(2):341-6. doi: 10.1093/humrep/17.2.341. PMID 11821275
- [Background] Coroleu B, Barri PN, Carreras O, Martinez F, Veiga A, Balasch J. The usefulness of ultrasound guidance in frozen-thawed embryo transfer: a prospective randomized clinical trial. Hum Reprod. 2002 Nov;17(11):2885-90. doi: 10.1093/humrep/17.11.2885. PMID 12407044
- [Background] Coroleu B, Barri PN, Carreras O, Belil I, Buxaderas R, Veiga A, Balasch J. Effect of using an echogenic catheter for ultrasound-guided embryo transfer in an IVF programme: a prospective, randomized, controlled study. Hum Reprod. 2006 Jul;21(7):1809-15. doi: 10.1093/humrep/del045. Epub 2006 Mar 23. PMID 16556674
- [Background] Matorras R, Mendoza R, Exposito A, Rodriguez-Escudero FJ. Influence of the time interval between embryo catheter loading and discharging on the success of IVF. Hum Reprod. 2004 Sep;19(9):2027-30. doi: 10.1093/humrep/deh366. Epub 2004 Jun 10. PMID 15192071
- [Background] Neithardt AB, Segars JH, Hennessy S, James AN, McKeeby JL. Embryo afterloading: a refinement in embryo transfer technique that may increase clinical pregnancy. Fertil Steril. 2005 Mar;83(3):710-4. doi: 10.1016/j.fertnstert.2004.08.022. PMID 15749502
- See also: Related Info — http://www.dexeus.com